CLINICAL TRIAL: NCT07404111
Title: An Adaptive Phase 1/2 MulticenteR Study Evaluating the Safety, Tolerability, Pharmacokinetics and EfficaCy of VV-14305 Delivered Via PeribuLbAr Injection in Patients With Moderate to Severe Thyroid Eye Disease (the RECLAIM Study)
Brief Title: A Study of VV-14305 for the Treatment of Thyroid Eye Disease
Acronym: RECLAIM
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Kriya Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: KRIYA-586-101
Record Dates: First submitted 2025-10-24; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Thyroid Eye Disease (TED)
MeSH Terms: conditions — Graves Ophthalmopathy | interventions — salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (6):
- Part 1 Cohort 1, low dose (Experimental): A single low dose of VV-14305 will be administered. In addition, prednisone will be administered prior to and after VV-14305.
  Interventions: Genetic: VV-14305
- Part 1 Cohort 2, mid dose (Experimental): A single mid dose of VV-14305 will be administered. In addition, prednisone will be administered prior to and after VV-14305.
  Interventions: Genetic: VV-14305
- Part 1 Cohort 3, high dose (Experimental): A single high dose of VV-14305 will be administered. In addition, prednisone will be administered prior to and after VV-14305.
  Interventions: Genetic: VV-14305
- Part 1 Optional Cohort 4, Part 2 dose (Experimental): A single dose of VV-14305 determined from Cohorts 1, 2, and 3 will be administered. In addition, prednisone will be administered prior to and after VV-14305.
  Interventions: Genetic: VV-14305
- Part 2 Treatment Arm (Experimental): A single dose of VV-14305 determined from Cohorts 1, 2, and 3 will be administered. In addition, prednisone will be administered prior to and after VV-14305.
  Interventions: Genetic: VV-14305
- Part 2 Sham Arm (Sham Comparator): A single sham injection will be administered. In addition, prednisone will be administered prior to and after the sham injection.
  Interventions: Other: Sham (No Treatment)

INTERVENTIONS:
Genetic: VV-14305 — VV-14305 will be administered via peribulbar injection.
  Arms: Part 1 Cohort 1, low dose; Part 1 Cohort 2, mid dose; Part 1 Cohort 3, high dose; Part 1 Optional Cohort 4, Part 2 dose; Part 2 Treatment Arm
Other: Sham (No Treatment) — Sham solution such as Saline
  Arms: Part 2 Sham Arm

SUMMARY:
The goal of this study is to evaluate the safety, tolerability, and efficacy of KRIYA-586 (VV-14305) in treating thyroid eye disease (TED).

ELIGIBILITY:
Inclusion Criteria:

1. Must be 18 to 80 years of age (inclusive) at Screening.
2. Body Mass Index (BMI) of 19 to 34 kg/m2 (inclusive).
3. Must be euthyroid (defined as normal thyroid-stimulating hormone) or have mild hyper- or hypothyroidism (being managed to bring them to a euthyroid state).
4. Best Corrected Visual Acuity (BCVA) score of 20/60 or better at Screening with no history of deterioration noted in the 3 months prior to Screening.
5. Must be willing and able to cease product use prior to VV-14305 (or sham) peribulbar injection if using non-steroidal anti-inflammatory drug (NSAIDs), medications or any herbal supplements, vitamins, or multivitamins with antiplatelet/anticoagulant properties.
6. The study eye and the fellow eye must fall within the pre-defined degree of proptosis and clinical activity score (CAS) as measured at Screening.
7. Participants must be diagnosed with TED prior to Screening and be diagnosed with Graves' disease and progressive moderate to severe TED at Screening.

Exclusion Criteria:

1. History of serious ocular condition(s) other than TED, including but not limited to uveitis, dry age-related macular degeneration (AMD), and wet AMD; Other orbital or ophthalmic diseases, including inflammatory conditions, optic neuropathy, tumors, glaucoma with visual field defect or visual field loss, that in the opinion of the Investigator and/or Medical Monitor is clinically significant.
2. Any medical, cognitive, or psychiatric condition that, in the opinion of the Investigator, could contraindicate the use of the investigational drug, make consistent study assessment and follow-up over the 12-month Post-Treatment Follow-up Period unlikely, or would make the participant an unsafe study candidate.
3. Diagnosed with diabetes (HbA1c ≥6.5%).
4. History of malignancy requiring chemotherapy and/or radiation in the 12 months prior to Screening, except for successfully treated nonmelanoma skin cancers (e.g., basal cell, squamous cell carcinomas), cervical intraepithelial neoplasia, and localized prostate cancer.
5. Known allergy or condition that would contraindicate the use of required study medications.
6. Any Screening assessment or laboratory value that, in the opinion of the Investigator and/or Medical Monitor, is clinically significant and renders the subject not suitable for study participation.
7. Any vaccination or planned vaccination 30 days prior to dosing, 4 weeks post dosing or during period of immunosuppression.
8. Participant requires or, in the opinion of the Investigator, is likely to require immediate surgical ophthalmological/orbital intervention or irradiation of either eye; Has had any prior surgery for TED including orbital decompression, strabismus surgery and any eyelid surgery on either eye.
9. Prior participation in other gene therapy, investigational drug, biologic or device clinical trials within 30 days prior to Screening.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2028-02 (Estimated); Study Completion 2029-02 (Estimated)

PRIMARY OUTCOMES:
Part 1: Safety and Tolerability of VV-14305 in participants with TED | 52 Weeks
  Incidence and severity of ocular and non-ocular adverse events, clinical laboratory values, physical examinations, vital signs, and ophthalmic examinations
Part 2: Safety of VV-14305 in Participants with TED Compared to Sham | 36 Weeks
  Incidence and severity of ocular and non-ocular adverse events, clinical laboratory values, physical examinations, vital signs, and ophthalmic examinations
Part 2: Efficacy of VV-14305 in participants with TED compared to Sham | 36 Weeks
  Percentage of participants with reduction in proptosis in the study eye as measured by exophthalmometer

SECONDARY OUTCOMES:
Part 1: Efficacy associated with VV-14305 in participants with TED | 52 Weeks
  Percentage of participants with reduction in proptosis in the study eye as measured by exophthalmometer
Efficacy associated with VV-14305 in participants with TED (as compared to Sham for Part 2) | 52 Weeks
  Percentage of participants with Baseline diplopia >0 who have a ≥1 grade reduction
Efficacy associated with VV-14305 in participants with TED (as compared to Sham for Part 2) | 52 Weeks
  Mean change from Baseline in extraocular muscle (EOM) volume within the study eye
Efficacy associated with VV-14305 in participants with TED (as compared to Sham for Part 2) | 52 Weeks
  Mean change from Baseline in EOM inflammation within the study eye
Efficacy associated with VV-14305 in participants with TED (as compared to Sham for Part 2) | 52 Weeks
  Mean change from Baseline in orbital fat volume (FV) within the study eye
Efficacy associated with VV-14305 in participants with TED (as compared to Sham for Part 2) | 52 Weeks
  Percentage of participants with a Clinical Activity Score (CAS) of 0 or 1 in the study eye
Effect of VV-14305 on quality of life (as compared to Sham for Part 2) | 52 Weeks
  Mean change from Baseline in overall score in the Graves Orbitopathy Quality of Life (GO-QoL) questionnaire, which includes two subscales: Visual Functioning and Appearance (scale range 0-100), where higher scores indicate better quality of life
Pharmacokinetics (PK) of VV-14305 transgene product | 52 Weeks
  Peak and steady-state concentrations of adeno-associated virus (AAV) vector-mediated transgene product in serum

CONTACTS AND LOCATIONS:
Locations (1):
- Kriya Clinical Trial Site, Auckland, New Zealand, New Zealand

IPD SHARING:
Plan to Share IPD: No